CLINICAL TRIAL: NCT05054023
Title: Randomized Clinical Trial of Topical Piroxicam Versus a New Herbal Medicine Based Gel in the Treatment of Acute Extremity Pain After Emergency Department Discharge
Brief Title: Topical Piroxicam vs Soulagel in the Treatment of Acute Extremity Pain After Emergency Department Discharge
Acronym: TPS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Monastir Emergency department, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Topic analgesics
Record Dates: First submitted 2021-09-10; First posted 2021-09-23 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Acute Pain
Keywords: soft tissues; trauma; topical; NSAID; herbal analgesics
MeSH Terms: conditions — Acute Pain; Wounds and Injuries | interventions — Piroxicam

STUDY DESIGN:
Intervention Model Description: The Soulagel was supplied in 50 ml tubes that contained rosemary essential oil (Romarinus offienalus), mint essential oil, clove essential oil (Eugenda caryophyllus), harpgophytum natural extract (Harpagophytum procumbens), meadowsweet natural extract (Filipendula ulmaria), aqua, methyl salicylate, menthol, camphre, carbomer, triethanolamine, polysorbate-20, sodium polyacrylate, trideceth-6, methylchloroisothiazolinone, methylisothiazolinone , magnesim Chloride and magnesium nitrater (Soulagel®; Belpharma Tunisia). Piroxicam gel was supplied in 50g tubes that contained 0.5% piroxicam.
  Study treatments were applied on the injured site3 times per day for 7 days. The gel must be gently rubbed on the skin over the injured site for 2 minutes.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization was performed centrally according to a computer-generated random list performed by a blinded study investigator who was not involved in any other part of the trial.
  All protocol treatments were administered in opaque tube with identical appearances and were numbered according to the randomization sequence by an independent nurse who was not involved in monitoring or follow-up of the subjects.
  the outcome assessor was also blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Piroxicam gel (Active Comparator): 50g tubes that contained 0.5% piroxicam. the gel was gently massaged in the injured site for 1 minute, 3 times a day for 7 days.
  Interventions: Drug: Arthrosyl®
- Soulagel®; Belpharma Tunisia (Active Comparator): 50 ml tubes that contained rosemary essential oil (Romarinus offienalus), mint essential oil, clove essential oil (Eugenda caryophyllus), harpgophytum natural extract (Harpagophytum procumbens), meadowsweet natural extract (Filipendula ulmaria), aqua, methyl salicylate, menthol, camphre, carbomer, triethanolamine, polysorbate-20, sodium polyacrylate, trideceth-6, methylchloroisothiazolinone, methylisothiazolinone , magnesim Chloride and magnesium nitrate. the gel was gently massaged in the injured site for 1 minute, 3 times a day for 7 days.
  Interventions: Drug: Soulagel®

INTERVENTIONS:
Drug: Soulagel® — topic gel
  Arms: Soulagel®; Belpharma Tunisia
Drug: Arthrosyl® — topic gel
  Other Names: piroxicam
  Arms: Piroxicam gel

SUMMARY:
Acute soft tissues injuries are a common complaint for emergency department (ED) visit. RICE and Topical non-steroidal anti-inflammatory drugs (NSAIDs) are frequently used to reduce pain and inflammation. Herbal therapy is commonly used to treat pain but few studies assessed its efficacy and tolerability.

DETAILED DESCRIPTION:
Materials and methods :

Study design It is a randomized, prospective, double blind, controlled, multicentric trial.

Study setting and selection of participants :

The trial is conducted in three community teaching hospitals :

* Emergency department, fattouma bourgiba university hospital, monastir, tunisia.
* Emergency department, sahloul university hospital, sousse, tunisia.
* Emergency department, farhat hached university hospital, sousse, tunisia.

The study includes patients aged 18 to 60 years who presented to the ED with acute soft-tissues limb trauma pain occurring within 24 hours before presentation, with a visual numeric scale (VNS) of 5 or more on a standard 11 point (0-10) and who required a prescription for home use analgesic treatment upon discharge. An informed consent is necessary. Pain was considered traumatic if it is reported as appearing immediately after the trauma.

Protocol :

After medical evaluation, every patient who meet the inclusion criteria, will receive randomly either Piroxicam gel or Soulagel tubes as detailed above according to the predetermined randomization.

None of the treating physician or nurses are aware about the medication received.

Adhesive and/or immobilizing casts, bandages, splints, and treatment by rest, ice, compression, or elevation were prohibited after randomization.

Patients could not take additional medications such as oral NSAIDs, opioids, muscle relaxants, or supplemental topical therapies.

Patients were phonelly contacted in order to ensure treatment adherence and evaluate VAS once a day until the end of the treatment. After the end of the treatment, patients' satisfaction with the treatment was noted and quoted as "not satisfied", "satisfied", and "very satisfied".

Need for rescue analgesic treatment was noted as well as the dose and duration. All patients were encouraged to report all adverse events during the treatment period. S

All data recorded on data collection sheets, including sex, demographics, medical history, and vital signs, were entered into SPSS (version 20.0 ; IBM corps) by the research manager.

Patients's informed consent is obtained. The ethic commitee of our institution approved the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to the ED with acute non-penetrating minor soft tissues musculoskeletal limb trauma occurring within 24 hours before presentation, and who required a prescription for home use analgesic treatment upon discharge for pain-on-movement (POM) with intensity >50 on a visual numeric scale (VNS) on a standard 11 point (0-10).
* Pain was considered traumatic if it is reported as appearing immediately after the trauma and no anterior pain was described in the same limb.

Exclusion Criteria:

* Pregnancy/Breastfeeding
* Skin lesions (excessive dryness or redness of the skin, atopic dermatitis, and eczema) in the painful region
* Presence of wound, joint dislocation, or more than one injury
* Presence of a fracture
* Severe trauma (ISS > 16)
* Hospitalization or surgery, daily use of NSAIDs or other analgesia within 2 weeks
* Previous treatment with analgesia for the same injury
* History of previous adverse reaction or known allergy or hypersensitivity
* Physical, visual, or cognitive impairment (inability to use the VNS pain score)
* Refusal to consent or to communicate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1525 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Treatment success resolution of pain with decrease of VAS more than 50% comparing to initial value at 30 minutes following analgesia administration | at seven days post ED discharge
  resolution of pain with decrease of visual numeric scale (that range from 0: no pain to 10 :severe pain) more than 50% comparing to initial value
Occurence of severe adverse events | at seven days post ED discharge
  occurence of severe adverse events

SECONDARY OUTCOMES:
Pain resolution time | at seven days post ED discharge
  time between the start of the analgesic treatment and the one when VNS (that range from 0: no pain to 10 :severe pain) decreased to less than 3.
The need for rescue analgesia and | at seven days post ED discharge
  doses of morphine required to reach efficient analgesia
Patient Satisfaction | at seven days post ED discharge
  Satisfaction of patients evaluated with the likert score at the ED discharge. (at 120 minutes patients were asked to rate the severity of nasal irritation on a 1 to 10 ordinal scale anchored.

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (1):
- Nouira Samir, Monastir, Emergency Department Monastir, Tunisia 5000, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided